CLINICAL TRIAL: NCT05972512
Title: A Randomized, Double-Blind, Placebo-Controlled, Safety, and Efficacy Study of Plant Based Biotin and Plant Based Biotin with Silica in Healthy Adult Human Subjects with Complaints of Hair Fall Thin, Dry, & Brittle Hair, and Dry Skin
Brief Title: A Clinical Study to Assess the Safety and Effectiveness of Plant-based Biotin and Plant Based Biotin with Silica in Healthy Human Subjects with Complaints of Hair Fall, Thin, Dry, & Brittle Hair, and Dry Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Orgenetics, Inc. (Industry)
Responsible Party: Principal Investigator, Dr Nayan Patel, Principal Investigator- Medical Director, NovoBliss Research Pvt Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NB230019-OI
Record Dates: First submitted 2023-07-07; First posted 2023-08-02 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2023-11

CONDITIONS: Hair Falling; Thin Hair; Dry Hair; Brittle Hair; Dry Skin
MeSH Terms: conditions — Alopecia | interventions — Silicon Dioxide

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-Blind, Placebo-Controlled, Safety, and Efficacy Study
Who Masked: Participant, Investigator
Masking Description: The study is double blind wherein neither the subjects nor the Investigator shall be aware of the test treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): The test treatment will be taken two times a day.
  Interventions: Other: Placebo
- Botanical Extract of standardised for biotin (1250 mcg) (Experimental): The standardised botanical extract of biotin is specially formulated for healthier hair and skin. Biotin promotes the hair growth.
  Interventions: Dietary Supplement: Botanical extract of standardized biotin
- Botanical Extract of standardised for biotin (1250mcg) + 10 mg Silica (Experimental): The standardised botanical extract of biotin and silica is specially formulated for healthier hair. The combination of biotin and silica will helpful in hair growth, reduces shedding, and improves the health of hair.
  Interventions: Dietary Supplement: Botanical extract of standardised biotin with silica

INTERVENTIONS:
Other: Placebo — Mode of usage: Two times a day Route of administration: Oral
  Arms: Placebo
Dietary Supplement: Botanical extract of standardized biotin — Mode of usage: Two times a day Route of administration: Oral
  Arms: Botanical Extract of standardised for biotin (1250 mcg)
Dietary Supplement: Botanical extract of standardised biotin with silica — Mode of usage: Two times a day Route of administration: Oral
  Arms: Botanical Extract of standardised for biotin (1250mcg) + 10 mg Silica

SUMMARY:
A randomized, double-blind, three-arm, placebo-controlled, safety, and efficacy study of plant-based Biotin and plant-based Biotin with Silica in healthy adult human subjects with complaints of hair fall, thin, dry, and brittle hair, and dry skin.

A sufficient number (maximum of 105 (35 subject/test treatment)) of female/male adult subjects will be recruited/enrolled to ensure a total of 96 subjects (32 subjects/test treatment) complete the study.

DETAILED DESCRIPTION:
The potential subjects will be screened as per the inclusion & exclusion criteria only after obtaining written informed consent from the subjects. Total study visits will be 8 during this study.

Visit 01 (Within 30 Days): Screening procedure, Informed consent obtain process, baseline evaluations, blood collection, tattoo on scalp, hair growth rate measurement Visit 02 (Day 01): Enrolments, hair growth rate measurement, other evaluations, product distribution, diary distribution, AE reporting (if any.

Visit 03 (Day 27 +2 Days): Treatment period, evaluations, tattoo, hair growth rate measurement, diary card review, AE reporting (if any).

Visit 04 (3 Days from Visit 03): Treatment period, evaluations, diary card review, AE Reporting (if any).

Visit 05 (Day 57 + 2Days): Treatment period, evaluations, tattoo, hair growth rate measurement, diary card review, AE Reporting (if any).

Visit 06 (3 Days from Visit 05): Treatment period, evaluations, diary card review, AE Reporting (if any).

Visit 07 (Day 87 +2 Days): Treatment period, evaluations, tattoo, hair growth rate measurement, diary card review, AE Reporting (if any).

Visit 08 (3 days from Visit 08): Evaluations, dairy card collection, AE reporting, test treatments accountability, End of Study process.

done on Day 04 before Day 01, Day 01 and after test treatment usage will be done on Day 27, Day 30, Day 57, Day 60, Day 87, Day 90 as listed-below.

* 60-S Hair Combing Method: Hair Fall.
* CASALite Nova (Phototrichogram): Hair Density, Thickness, Hair Growth Rate, Scalp Condition.
* PGA Score: Signs of brittle nails, surface roughness, raggedness and peeling.
* Visioscan®VC 20plus (C+K Instrument): Crow's feet area wrinkles, fine lines, skin texture - roughness, dryness, wrinkles, smoothness (Right cheek).
* MoitureMeterEPiD: Skin hydration (Right cheek).
* Hair Pull Test: Hair strength.
* Pluck Test: A:T ratio (Hair Growth Cycle)
* Cutometer: Skin elasticity (Right cheek).
* PGA Griffith Scale: Skin dryness, redness, fine wrinkling/lines, coarse wrinkling/lines, laxity, roughness and sallowness
* Tewameter® TM 300: Skin barrier function (Right Cheek)
* General Appearance of Hair: Hair shininess, hair reflection, hair plasticity, hair fizziness, hair volume, hair density Digital photographs: Facial photographs before test treatment consumption and after test treatment consumption
* Blood parameters: CBC, total Serum Cholesterol, Triglyceride, Random Glucose, LDL, HDL [Note: blood collection will be performed on Day 01 And Day 90]
* Blood parameter: HBsAg (Hepatitis B surface antigen) - Screening only
* Subjective product perception assessment regarding the test treatment's effect on skin elasticity, suppleness, skin color, fragrance, taste, skin hydration, skin tone, firmness, appearance, hair and nails, strongness and shine.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20 to 60 years (both inclusive) at the time of consent
2. Sex: Healthy males and non-pregnant/non-lactating females.
3. Subject have complaints of hair fall, thin, dry and brittle hair, and dry skin.
4. Females of childbearing potential must have a reported negative pregnancy test.
5. Subject are generally in good health.
6. Subject must have negative Hepatitis B Surface Antigen Test at baseline.
7. Subject with self-proclaimed nonpathological thin, dry and brittle hair.
8. Subject is willing to forgo cosmetic procedures 3 months prior to and for the duration of the study.
9. Subject is able to remain on stable doses of contraceptive or replacement hormonal therapy, including no therapy, 6 weeks prior to and for the duration of the study.
10. Subject is able to follow their normal skin care routines and to refrain from introducing any new skin care products during the study.
11. Subject is able to forgo changes in baseline medications and nutritional supplements during the study period.
12. If the subject is of childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post-menopausal for at least 1 year or have had a tubal ligation.
13. If currently using hormonal contraception, has been using this form of contraception for at least 6 months and agrees to continue using the same contraception for the duration of the study.
14. Subjects are willing not to introduce any new soaps, cleansers, laundry detergents, lotions, creams, shampoos etc. for the duration of the study.
15. Subjects are willing to give written informed consent and are willing to follow the study procedure.
16. Subjects who have used other marketed products for hair thinning in the past.
17. Subjects who commit not to use medicated/ prescription shampoos/hair care products (containing Minoxidil / Anti-thinning agents) or any other hair growth, treatment for thin hair, or hair products other than the test treatments for the entire duration of the study.
18. Willing to use test treatments throughout the study period.

Exclusion Criteria:

1. Subjects with a history of hair thinning/hair fall due to any clinically significant self-reported problems/s like anaemia, thyroid problems, etc.
2. Subject has a history of allergy or sensitivity to the test treatment ingredients.
3. Subject has a history of any dermatological condition of the scalp other than hair loss and/or dandruff or active dermatological condition that might interfere with the clinical assessments (e.g. tattoos, eczema, psoriasis, acne, etc.).
4. Subject has used any systemic therapy with chronic antibiotic therapy, retinoids, and/or oral steroids during the 4 weeks prior to the start or anticipates having to use at any point during the study.
5. Subject has applied any topical retinoids within 2 weeks of the screening visit or anticipates having to use at any point during the study.
6. Subject is not willing to avoid unprotected sun or other UV radiation exposure during the study period.
7. Subject is currently pregnant/breastfeeding.
8. Subject has a history of prior use of hair growth treatment within 3 months.
9. Subject has a history of any prior hair growth procedures (e.g., hair transplant or laser).
10. Subject has a history of alcohol or drug addiction.
11. Subjects who have plans of shaving scalp hair during the study.
12. Subject has a past or present condition of irritated or visibly inflamed scalp or severe scalp disease.
13. Any other condition which could warrant exclusion from the study, as per the dermatologist's/investigator's discretion.
14. Pregnant or breastfeeding or planning to become pregnant during the study period.
15. History of chronic illness which may influence the cutaneous state.
16. Subjects participating in other similar nutraceuticals, food, supplemental or therapeutic trials or hair/scalp/skin care products within the last four weeks.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Change in hair fall | Baseline (Day 01) before dosing to Day 30, Day 60, Day 90 post-dose, between treatments, within treatment and compare with placebo arm
  To assess the effectiveness of test treatment in terms of change in hair fall by using 60-s hair comb test
Change in hair thickness (Unit= µm) | From baseline (Day 01) before dosing to Day 30, Day 60 and Day 90 post-dose, between treatments, within treatment and compare with placebo arm
  To assess the effectiveness of test treatment in terms of change in hair thickness by CASALite Nova thorough Phototrichogram
Change in hair growth rate (Unit= µm) | From screening (Within 4 Day) to Day 01, Day 27, Day 30, Day 57, Day 60, Day 87 and Day 90 post-dose, between treatment, within treatment, and compare with placebo arm
  To assess the effectiveness of test treatment in terms of change in hair growth rate by using CASALite Nova thorough Phototrichogram
Change in PGA score for sign of brittle nails | Baseline (Day 01) before dosing of test treatments to Day 30, Day 60 and Day 90 post-dose, between treatments, within treatment and compare with placebo treated arm
  To assess the effectiveness of test treatment in terms of change in PGA score for sign of brittle nails by using 5-point scoring scale Where 0= None and 5= Severe
Change in Hair Density (Unit= sqcm) | rom baseline (Day 01) before dosing to Day 30, Day 60 and Day 90 post-dose, between treatments, within treatment and compare with placebo arm
  o assess the effectiveness of test treatment in terms of change in hair density by using CASALite Nova thorough phototrichogram
Change in PGA score for sign of Nail Surface Roughness | From baseline (Day 01) before dosing of test treatments to Day 30, Day 60 and Day 90 post-dose, between treatments, within treatment and compare with placebo treated arm
  To assess the effectiveness of test treatment in terms of change in PGA score for sign of nail surface roughness by using 3 point scoring scale Where 0= None, 3= Severe
Change in PGA score for sign of Surface Raggedness | From baseline (Day 01) before dosing of test treatments to Day 30, Day 60 and Day 90 post-dose, between treatments, within treatment and compare with placebo treated arm
  To assess the effectiveness of test treatment in terms of change in PGA score for sign of nail surface raggedness by using 3 point scoring scale Where 0= None, 3= Severe
Change in PGA score for sign of Peeling | From baseline (Day 01) before dosing of test treatments to Day 30, Day 60 and Day 90 post-dose, between treatments, within treatment and compare with placebo treated arm
  To assess the effectiveness of test treatment in terms of change in PGA score for sign of nail surface peeling by using 4 point scoring scale where 0= none, 3= severe

SECONDARY OUTCOMES:
Change in facial wrinkle | From baseline (Day01) to Day 30, Day 60 and Day 90, between treatments, within treatment and compare with placebo treated arm
  To assess the effectiveness of test treatment in terms of change in facial wrinkles by using Visioscan VC 20plus (Instrumental Evaluation)
Change in fine lines of crow's feet area, | from baseline (Day01) to Day 30, Day 60 and Day 90, between treatments, within treatment and compare with placebo treated arm
  To assess the effectiveness of test treatment in terms of change in fine lines of crow's feet area by using Visioscan VC 20plus (Instrumental Evaluation)
Change in skin hydration | from baseline (Day01) to Day 30, Day 60 and Day 90, between treatments, within treatment and compare with placebo treated arm
  To assess the effectiveness of test treatment in terms of change in skin hydration by using MoistureMeterEpiD (Instrumental Evaluation)
Change in hair Strength | From baseline (Day01) before dosing to Day 30, Day 60 and Day 90 post-dose, between treatments, within treatment and compare with placebo treated arm
  To assess the effectiveness of test treatment in terms of change in hair strength by using hair pull test
Change in skin elasticity | From baseline (Day01) before dosing to Day 30, Day 60 and Day 90 post-dose, between treatments, within treatment and compare with placebo treated arm
  To assess the effectiveness of test treatment in terms of change in skin elasticity by using Cutometer Dual MPA 580(Instrumental Evaluation)
Change in PGA Score | From baseline (Day01) before dosing to Day 30, Day 60 and Day 90 post-dose, between treatments, within treatment and compare with placebo treated arm
  To assess the effectiveness of test treatment in terms of change in PGA scores i.e. dryness, redness, fine lines, coarse wrinkle, laxity, roughness, and sallowness by using Griffith scale Where 0= No appearance and 9= Severe
Change in barrier function of skin | From baseline (Day01) before dosing to Day 30, Day 60 and Day 90 post-dose, between treatments, within treatment and compare with placebo treated arm
  To assess the effectiveness of test treatment in terms of change in barrier function of skin by using Tewameter TM Hex(Instrumental Evaluation)
Change in general appearance of hair | From baseline (Day01) before dosing to Day 30, Day 60 and Day 90 post-dose, between treatments, within treatment and compare with placebo treated arm
  To assess the effectiveness of test treatment in terms of change in general appearance of hair such as hair shininess, hair reflection, hair volume, hair density, hair plasticity, hair frizziness by dermatologist trained evaluator
Change in Anagen: Telogen ratio | From baseline (Day01) to Day 90 (+2Days), between treatments, within treatment and compare with placebo treated arm
  To assess the effectiveness of test treatment in terms of change in Anagen: Telogen ratio of hair by using hair pluck test
Change in facial photographs(Left/Center/Right) | From baseline before usage of test treatments on Day 01, and after usage of test treatments on Day 30, Day 60, Day 90
  Change in facial photographs (Left/Center/Right) of the subject by using Nikol Digital Camera D3300
Treatment perception questionnaire | From before dosing of test treatments to after usage of test treatments on Day 30, Day 60, Day 90
  To assess the effectiveness of test treatment in terms of treatment perception by using 9 point hedonic scale
Change in Complete Blood Count | From Day 01 and Day 90
  Safety of test treatment will be assessed in terms of difference in Complete Blood Count
Change in silicon deposits on hair cuticle | From baseline (Day01) before dosing to Day 90 post-dose, between treatments, within treatment and compare with placebo treated arm
  To assess the effect of test treatments in terms of change silicon deposits on hair cuticle by using Scanning Electrone Microscope (8 subject/ test treatment)
Change in Skin Texture | From baseline (Day01) to Day 30, Day 60 and Day 90, between treatments, within treatment and compare with placebo treated arm
  To assess the effectiveness of test treatment in terms of change in Skin texture by using Visioscan VC 20plus
Change in Total Serum Cholesterol | From Day 01 and Day 90
  Safety of test treatment will be assessed in terms of difference in Total Serum Cholesterol level
Change in Triglycerides | From Day 01 and Day 90
  Safety of test treatment will be assessed in terms of difference in Triglycerides level
Change in LDL level | From Day 01 and Day 90
  Safety of test treatment will be assessed in terms of difference in LDL level
Change in HDL level | From Day 01 and Day 90
  Safety of test treatment will be assessed in terms of difference in HDL level
Change in Random Glucose Level | From Day 01 and Day 90
  Safety of test treatment will be assessed in terms of difference in Random Glucose Level

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nayan K Patel, Principal Investigator — Medical Direcor
Locations (1):
- NovoBliss Research Pvt Ltd, Gandhinagar, Gujarat, India

IPD SHARING:
Plan to Share IPD: No